CLINICAL TRIAL: NCT01531075
Title: Assessment of Hepatitis B Vaccination Efficacy in Patients With Inflammatory Bowel Diseases
Brief Title: Hepatitis B Vaccine in Patients With Inflammatory Bowel Disease
Acronym: HBV VIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Ohad Etzion, Senior physician, Department of Gastroenterology and Liver Disease, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: sor026511ctil
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Inflammatory Bowel Disease
Keywords: HBV, Inflammatory bowel disease, immunosuppressor
MeSH Terms: conditions — Inflammatory Bowel Diseases; Hepatitis B | interventions — Engerix-B; Pre-S vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ENGERIX-B (Experimental)
  Interventions: Biological: ENGERIX-B (HBV Vaccine)
- Sci-B-Vac (Experimental)
  Interventions: Biological: Sci-B-Vac

INTERVENTIONS:
Biological: ENGERIX-B (HBV Vaccine) — ENGERIX-B (Hepatitis B Vaccine) 20 mcg, A series of 3 doses (1 mL each) given on a 0-, 1-, 6-month schedule.
  Other Names: ENGERIX-B
  Arms: ENGERIX-B
Biological: Sci-B-Vac — Sci-B-Vac (Hepatitis B Vaccine) 10 μg/ml, A series of 3 doses (1 mL each) given on a 0-, 1-, 6-month schedule.
  Arms: Sci-B-Vac

SUMMARY:
The objective is to assess the efficacy of Hepatitis B Virus vaccination in a population of IBD patients treated with immunosuppressive medications.

ELIGIBILITY:
Inclusion Criteria:

* Male/female ≥ 18 years of age
* Evidence of IBD as diagnosed by clinical, laboratory imaging and endoscopic criteria.
* Treated with at least one immunosuppressive medication at the time of study initiation
* Provided written informed consent.

Exclusion Criteria:

* Pregnant women
* Diagnosis of chronic viral hepatitis B
* Any major acute medical event in the 30 days prior to recruitment that necessitated hospitalization ( acute myocardial infarction, CVA, pulmonary emboli, sepsis, major trauma)
* Any other chronic inflammatory condition not related to IBD ( connective tissue disease, Chronic liver disease, COPD, poorly controlled diabetes mellitus)
* Active hematologic or oncologic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
protective level of anti HBs antibodies | 1 month after the last does of vaccine
  Antibody titer >10 IU/ml 30 days following last vaccine dose will be considered protective.
  In the work done by Altunoz et al., titer rate below 10 IU was observed in 40% of the patients, while 40% of the patients achieved a rate of above 100 IU. Therefore, we can estimate that the geometric mean of distribution is approx. 50 IU. A sample size of 37 patients in each group achieves a power of 80% to detect a ratio above 1.37 between the two vaccinated groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Etzion, MD, Principal Investigator — Soroka UMC
Locations (1):
- Soroka UMC, Beersheba, Israel